CLINICAL TRIAL: NCT01607190
Title: Biomarkers of Diabetic Retinopathy Progression.
Acronym: C-Tracer
Status: Completed | Type: Observational
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Responsible Party: Sponsor
Other Study IDs: 4C-2012-02
Record Dates: First submitted 2012-05-23; First posted 2012-05-30 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Type 2 Diabetes Mellitus; Mild Nonproliferative Diabetic Retinopathy
Keywords: type 2 diabetes mellitus; nonproliferative diabetic retinopathy
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with diabetic retinopathy.

SUMMARY:
The purpose of this study is to validate a predictive model of diabetic retinopathy progression in patients with diabetes mellitus type 2 patients to clinically significant macular edema (CSME) needing treatment either photocoagulation or intravitreal injections (ITV) using non-invasive techniques.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Age over 35 years-old
* Non-proliferative diabetic retinopathy (Levels 20 to 35, according the ETDRS criteria)
* Best Corrected Visual Acuity > 20/25 on the ETDRS chart
* Informed Consent

Exclusion Criteria:

* Previous laser therapy
* Other retinal vascular disease
* Glaucoma
* Recent intraocular surgery (in the last 6 months)
* Inadequate ocular media and/ or pupil dilatation that do not permit good quality fundus photography (e.g. cataract)
* HbA1C > 11 % at the Screening
* Subject that has a condition or that is in a situation which may put him/her at significant risk, may confound the study results or may interfere significantly with his/ her participation in the study.

Ages: 35 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes mellitus and mild nonproliferative diabetic retinopathy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-11; Primary Completion 2016-04 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
CSME needing treatment either photocoagulation or ITV. | Months 0, 6, 12 and 24.

SECONDARY OUTCOMES:
Best corrected visual acuity. | Months 0, 6, 12 and 24.
Vision loss of at least 2 lines documented in ETDRS charts | Months 0, 6, 12 and 24.
Central retinal thickness | Months 0, 6, 12 and 24.
Microaneurysm(MA) activity (number of MA, MA formation and MA disappearance rates and MA turnover) | Months 0, 6, 12 and 24.

CONTACTS AND LOCATIONS:
Overall Officials: José Cunha-Vaz, MD, PhD, Study Chair — Association for Innovation and Biomedical Research on Light and Image
Locations (2):
- LV Prasad Eye Institute, Hyderabad, Andhra Pradesh, India
- AIBILI- Association for Biomedical Research and Inovation on Light and Image., Coimbra, Portugal

REFERENCES:
- [Derived] Cunha-Vaz J, Ribeiro L, Costa M, Simo R. Diabetic Retinopathy Phenotypes of Progression to Macular Edema: Pooled Analysis From Independent Longitudinal Studies of up to 2 Years' Duration. Invest Ophthalmol Vis Sci. 2017 May 1;58(6):BIO206-BIO210. doi: 10.1167/iovs.17-21780. PMID 28785768